CLINICAL TRIAL: NCT01857687
Title: Noninvasive Evaluation of Ischemia Causing Coronary Stenosis, Wall Shear Stress, and Total Plaque Force Using Coronary CT Angiography (CCTA) and Physics-based Analytic Model Derived From Conservation of Energy
Brief Title: Evaluation of FFR, WSS, and TPF Using CCTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate Professor of Medicine / Cardiology, Seoul National University Hospital
Other Study IDs: SNUH CT-FFR WSS TPF
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: To Assess the Feasibility of CT-derived FFR, WSS and TPF on Coronary Atherosclerotic Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients with coronary artery stenosis

SUMMARY:
To assess the feasibility of CT-derived computed fractional flow reserve (FFRCT), wall shear stress and total plaque force on coronary atherosclerotic plaque and to collect the preliminary data to apply those parameters for the prediction of clinical outcomes in patients with coronary artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with available CCTA within 3 months of invasive angiography and invasive imaging methods (IVUS or OCT)

Exclusion Criteria:

* Poor CT images (unable to reconstruct 3 dimensional coronary artery model)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coronary artery stenosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
CT-derived computed fractional flow reserve | at time of evaulation

SECONDARY OUTCOMES:
wall shear stress | at time of evaulation
total plaque force | at time of evaulation

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University hospital, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Fearon WF, Bornschein B, Tonino PA, Gothe RM, Bruyne BD, Pijls NH, Siebert U; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) Study Investigators. Economic evaluation of fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. Circulation. 2010 Dec 14;122(24):2545-50. doi: 10.1161/CIRCULATIONAHA.109.925396. Epub 2010 Nov 29. PMID 21126973
- [Background] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493
- [Background] Wong JT, Le H, Suh WM, Chalyan DA, Mehraien T, Kern MJ, Kassab GS, Molloi S. Quantification of fractional flow reserve based on angiographic image data. Int J Cardiovasc Imaging. 2012 Jan;28(1):13-22. doi: 10.1007/s10554-010-9767-0. Epub 2011 Jan 7. PMID 21213051
- [Background] Hamon M, Biondi-Zoccai GG, Malagutti P, Agostoni P, Morello R, Valgimigli M, Hamon M. Diagnostic performance of multislice spiral computed tomography of coronary arteries as compared with conventional invasive coronary angiography: a meta-analysis. J Am Coll Cardiol. 2006 Nov 7;48(9):1896-910. doi: 10.1016/j.jacc.2006.08.028. Epub 2006 Sep 26. PMID 17084268
- [Background] Achenbach S, Moselewski F, Ropers D, Ferencik M, Hoffmann U, MacNeill B, Pohle K, Baum U, Anders K, Jang IK, Daniel WG, Brady TJ. Detection of calcified and noncalcified coronary atherosclerotic plaque by contrast-enhanced, submillimeter multidetector spiral computed tomography: a segment-based comparison with intravascular ultrasound. Circulation. 2004 Jan 6;109(1):14-7. doi: 10.1161/01.CIR.0000111517.69230.0F. Epub 2003 Dec 22. PMID 14691045
- [Background] Leber AW, Knez A, von Ziegler F, Becker A, Nikolaou K, Paul S, Wintersperger B, Reiser M, Becker CR, Steinbeck G, Boekstegers P. Quantification of obstructive and nonobstructive coronary lesions by 64-slice computed tomography: a comparative study with quantitative coronary angiography and intravascular ultrasound. J Am Coll Cardiol. 2005 Jul 5;46(1):147-54. doi: 10.1016/j.jacc.2005.03.071. PMID 15992649
- [Background] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Samady H, Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Maynard C, Timmins LH, Quyyumi AA, Giddens DP. Coronary artery wall shear stress is associated with progression and transformation of atherosclerotic plaque and arterial remodeling in patients with coronary artery disease. Circulation. 2011 Aug 16;124(7):779-88. doi: 10.1161/CIRCULATIONAHA.111.021824. Epub 2011 Jul 25. PMID 21788584
- [Background] Stone PH, Saito S, Takahashi S, Makita Y, Nakamura S, Kawasaki T, Takahashi A, Katsuki T, Nakamura S, Namiki A, Hirohata A, Matsumura T, Yamazaki S, Yokoi H, Tanaka S, Otsuji S, Yoshimachi F, Honye J, Harwood D, Reitman M, Coskun AU, Papafaklis MI, Feldman CL; PREDICTION Investigators. Prediction of progression of coronary artery disease and clinical outcomes using vascular profiling of endothelial shear stress and arterial plaque characteristics: the PREDICTION Study. Circulation. 2012 Jul 10;126(2):172-81. doi: 10.1161/CIRCULATIONAHA.112.096438. Epub 2012 Jun 21. PMID 22723305
- [Derived] Choi G, Lee JM, Kim HJ, Park JB, Sankaran S, Otake H, Doh JH, Nam CW, Shin ES, Taylor CA, Koo BK. Coronary Artery Axial Plaque Stress and its Relationship With Lesion Geometry: Application of Computational Fluid Dynamics to Coronary CT Angiography. JACC Cardiovasc Imaging. 2015 Oct;8(10):1156-1166. doi: 10.1016/j.jcmg.2015.04.024. Epub 2015 Sep 9. PMID 26363834